CLINICAL TRIAL: NCT00567307
Title: The Feasibility of a Polypill Clinical Trial for Primary Prevention of Cardiovascular Disease: A Pilot Study
Brief Title: Polypill For Prevention of Cardiovascular Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: World Health Organization (Other); National Hospital of Sri Lanka (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00004134; SLCTR/ 2007/012 (Registry Identifier: Sri Lanka IRB)
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- The Red Heart Pill 2b (Polypill) (A) (Experimental): The Polypill is composed of 75 mg aspirin, 20 mg simvastatin, 10 mg lisinopril and 12.5 mg hydrochlorothiazide
  Interventions: Drug: Red Heart Pill 2b (Polypill)
- Standard Practice Group (B) (Active Comparator): Standard Practice
  Interventions: Other: Standard Practice

INTERVENTIONS:
Drug: Red Heart Pill 2b (Polypill) — Arm A will receive the polypill (Red Heart pill 2b) which is a combination of aspirin (75 mg), simvastatin (20g), lisinopril (10mg) and hydrochlorothiazide (12.5 mg)
  Other Names: Polypill
  Arms: The Red Heart Pill 2b (Polypill) (A)
Other: Standard Practice — Arm B will receive management of their CVD risk according to the usual care given to participants in similar conditions
  Other Names: Usual care
  Arms: Standard Practice Group (B)

SUMMARY:
The purpose of this pilot study is to provide data on the feasibility of conducting a large clinical trial on the polypill (combination of aspirin, angiotensin converting enzyme inhibitor, thiazide diuretic, and statin) for primary prevention of cardiovascular disease (CVD). We hypothesized that A "polypill" comprising the aforementioned four components would significantly reduce the estimated 10-year total CVD risk score with high adherence and no significant increase in adverse effects compared to the standard practice.

DETAILED DESCRIPTION:
This is an open-label, parallel-group, randomized clinical trial comparing a Polypill to Standard Practice (defined as usual care administered to patients with similar conditions). Approximately 200 participants will be recruited from three sites in Sri Lanka: The National Hospital of Sri Lanka, Colombo; Teaching Hospital, Kegalle, and Teaching Hospital, Kandy. Subsequent to granting written informed consent, patients will undergo screening and baseline evaluation to confirm eligibility, followed by randomization to the Polypill or to the Standard Practice study arm. Patients receiving either intervention will return for a total of three monthly clinic visits.

Physician acceptability will be evaluated through a five-question survey will be mailed to a random sample of physicians from the participating clinical sites and to the Council of General Practitioners in Sri Lanka.

Patient acceptability will be measured in participants who will complete the study as well as those who will be screened but not eligible

ELIGIBILITY:
Inclusion Criteria:

* Estimated 10-year total CVD risk score > 20%. The total CVD risk assessment will be based on the recently developed WHO CVD risk prediction charts
* No contraindication for treatment with aspirin, angiotensin converting enzyme inhibitors, low-dose diuretics, or statins
* Informed consent given

Exclusion Criteria:

* Patients with established angina pectoris, coronary heart disease, myocardial infarction, transient ischemic attacks, stroke, peripheral vascular disease, coronary revascularization and/or carotid endarterectomy Left ventricular hypertrophy (on ECG) or hypertensive retinopathy (grade III or IV)
* Patients with secondary hypertension
* Patients with diabetes type 1 or 2 with overt neuropathy or other significant renal disease.
* Known renal failure or impairment
* Atrial fibrillation
* ALT > 1.5 times the upper limit of normal
* History of liver cirrhosis or hepatitis
* History of recent gastrointestinal bleeding (within the last year)
* Women in child bearing period
* History of life-limiting diseases or events
* Unwillingness to sign informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elsayed Z Soliman, MD, MSc, MS, Principal Investigator — Wake Forest University Health Sciences; Shanthi Mendis, MD, FRCP, Study Director — World Heath Organization; Curt D Furberg, MD, PhD, Study Chair — Wake Forest University Health Sciences
Locations (3):
- Sri Lanka (3):
  - The National Hospital of Sri Lanka, Colombo
  - Teaching (General) Hospital Kandy, Kandy
  - Teaching (General) Hospital Kegalle, Kegalle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soliman EZ, Mendis S, Dissanayake WP, Somasundaram NP, Gunaratne PS, Jayasingne IK, Furberg CD. A Polypill for primary prevention of cardiovascular disease: a feasibility study of the World Health Organization. Trials. 2011 Jan 5;12:3. doi: 10.1186/1745-6215-12-3. PMID 21205325

RESULTS

PARTICIPANT FLOW:
Groups:
- The Polypill Group (Arm A): The Polypill Group (Arm A) received a Polypill composed of 75 mg aspirin, 20 mg simvastatin, 10 mg lisinopril and 12.5 mg hydrochlorothiazide
  Red Heart Pill 2b (Polypill): Arm A will receive the polypill (Red Heart pill 2b) which is a combination of aspirin (75 mg), simvastatin (20g), lisinopril (10mg) and hydrochlorothiazide (12.5 mg)
- Standard Practice Group (Arm B): Standard Practice
  Standard Practice: Arm B received management of their CVD risk according to the usual care given to participants in similar conditions
Period: Overall Study
Arm/Group | The Polypill Group (Arm A) | Standard Practice Group (Arm B)
Started | 111 | 105
Completed | 99 | 104
Not Completed | 12 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Polypill Group (Arm A) | Standard Practice Group (Arm B) | Total
Number analyzed (Participants) | 111 | 105 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (7.4) | 59.0 (6.9) | 59.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 80 | 157
  Male | 34 | 25 | 59
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHG] | 164.7 (17.3) | 165.7 (19.2) | 165.2 (18.2)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.7 (1.3) | 6.1 (1.3) | 5.9 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Reduction of the Estimated 10-year Total Cardiovascular Risk Score
Description: Estimated 10-year CVD total risk score were calculated in the field centers and in the Coordinating Center from the measures of blood pressure and total cholesterol and from the medical history data collected during each visit using the WHO CVD prediction chart. The estimated 10-year CVD total risk calculated by the Coordinating Center were used for analysis. the score is based on systolic blood pressure and total cholesterol measures as well as on medical history data (monthly). Each one of these risk factors is assigned a point in the score and then linked to a table that mention the calculated CVD risk
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | The Polypill Group (Arm A) | Standard Practice Group (Arm B)
Number analyzed (Participants) | 99 | 104
percent | 11.5 (113.0) | 11.1 (10)

ADVERSE EVENTS:
Time Frame: Cumulative frequency of major side effects during the 3-month treatment period by study group among those who completed the study (99 in the polypill group and 104 in the standard practice)
Description: This is among those who completed the study (99 in the polypill group and 104 in the standard practice)
Arm/Group | The Polypill Group (Arm A) | Standard Practice Group (Arm B)
Serious Adverse Events (participants affected / at risk) | 26/99 | 29/104
Other Adverse Events (participants affected / at risk) | 15/99 | 12/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Polypill Group (Arm A) (N=99) | Standard Practice Group (Arm B) (N=104)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 26 (26) | 29 (29)
Epigastric pain (Gastrointestinal disorders) | 15 (15) | 20 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 18 (18)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Polypill Group (Arm A) (N=99) | Standard Practice Group (Arm B) (N=104)
Fatigue (General disorders) | 15 (15) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No